CLINICAL TRIAL: NCT01168934
Title: A Phase 1, Single Dose, Randomized, Cross-Over Absolute Bioavailability Study In Healthy Volunteers Comparing Oral To Intravenous Administration Of Crizotinib (PF-02341066)
Brief Title: A Phase 1 Absolute Bioavailability Study For Oral Crizotinib In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: A8081010
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Results first posted 2011-10-19 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: healthy volunteers; crizotinib; absolute bioavailability; pharmacokinetics
MeSH Terms: interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Each subject will receive single oral and IV doses of crizotinib separated by at least 14 days.
  Interventions: Drug: crizotinib

INTERVENTIONS:
Drug: crizotinib — Treatment A: Intravenous dose of 50 mg crizotinib will be administered as directed.
Drug: crizotinib — Treatment B: Oral dose of 250 mg crizotinib as 1 × 50-mg Immediate Release Tablet and 2 × 100-mg Immediate Release Tablets will be administered in the fasted state as directed.

SUMMARY:
This study will be an open-label, randomized, 2-period, 2-treatment, 2-sequence, cross-over single-dose study to test the absolute bioavailability of oral crizotinib formulation to IV formulation in healthy adult volunteers. Fourteen (14) subjects will be enrolled to obtain at least 12 evaluable subjects who complete the study. Each subject will receive two treatments (A and B) with a washout period of at least 14 days between each treatment.

DETAILED DESCRIPTION:
evaluate the absolute bioavailability of oral crizotinib to IV crizotinib.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female of non-childbearing potential subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m^2; and a total body weight >50 kg (110 lbs)

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males within 6 months of screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.
* 12-lead ECG demonstrating QTc >450 msec at Screening.
* Pregnant or nursing females; females of childbearing potential, including those with tubal ligation.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. Herbal supplements and hormone replacement therapy must be discontinued 28 days prior to the first dose of study medication.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* A positive serology for Hepatitis B or Hepatitis C.
* Subjects who are currently smoking.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081010&StudyName=A%20Phase%201%20Absolute%20Bioavailability%20Study%20For%20Oral%20Crizotinib%20In%20Healthy%20Volunteers

RESULTS

PARTICIPANT FLOW:
Groups:
- Crizotinib 50 mg IV First, Then Crizotinib 250 mg Oral: Single intravenous (IV) dose of crizotinib 50 milligram (mg) in first intervention period; and single oral dose of crizotinib 250 mg immediate release tablet (IRT) in second intervention period. A washout period of at least 14 days was maintained between each period.
- Crizotinib 250 mg Oral First, Then Crizotinib 50 mg IV: Single oral dose of crizotinib 250 mg IRT in first intervention period; and single IV dose of crizotinib 50 mg in second intervention period. A washout period of at least 14 days was maintained between each period.
Period: First Intervention Period
Arm/Group | Crizotinib 50 mg IV First, Then Crizotinib 250 mg Oral | Crizotinib 250 mg Oral First, Then Crizotinib 50 mg IV
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Washout Period (at Least 14 Days)
Arm/Group | Crizotinib 50 mg IV First, Then Crizotinib 250 mg Oral | Crizotinib 250 mg Oral First, Then Crizotinib 50 mg IV
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Second Intervention Period
Arm/Group | Crizotinib 50 mg IV First, Then Crizotinib 250 mg Oral | Crizotinib 250 mg Oral First, Then Crizotinib 50 mg IV
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes participants randomized to receive crizotinib 50 mg IV first and crizotinib 250 mg oral first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 35.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Dose Normalized Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC [0 - ∞][dn])
Description: AUC [0 - ∞][dn] = Dose normalized area under the plasma concentration versus time curve (AUC[dn]) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - ∞) divided by dose.
Time Frame: 0 (pre-dose), 1, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 144 hours (hrs) post IV crizotinib dose in Treatment A and 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, and 144 hrs post oral crizotinib dose in Treatment B
Population: Pharmacokinetic (PK) parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL/mg
Groups:
- Crizotinib 50 mg IV: Single IV dose of crizotinib 50 mg (Treatment A [Reference]) in either intervention period.
- Crizotinib 250 mg Oral: Single oral dose of crizotinib 250 mg (Treatment B [Test]) in either intervention period.
Arm/Group | Crizotinib 50 mg IV | Crizotinib 250 mg Oral
Number analyzed (Participants) | 14 | 14
ng*hr/mL/mg | 21.36 (3.99) | 9.28 (3.32)
Statistical Analysis 1: Comparison: Crizotinib 50 mg IV vs Crizotinib 250 mg Oral; Natural log transformed AUC (0 - ∞)(dn) of crizotinib was analyzed using mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% confidence intervals (CIs) for the differences was exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 43.44, 90% CI 2-sided [39.68 to 47.56]

2. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC [0 - ∞])
Description: AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: 0 (pre-dose), 1, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 144 hrs post IV crizotinib dose in Treatment A and 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, and 144 hrs post oral crizotinib dose in Treatment B
Population: PK parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib 50 mg IV | Crizotinib 250 mg Oral
Number analyzed (Participants) | 14 | 14
ng*hr/mL | 1067.00 (198.54) | 2321.00 (833.14)

3. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration (AUClast).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib 50 mg IV | Crizotinib 250 mg Oral
Number analyzed (Participants) | 14 | 14
ng*hr/mL | 1007.00 (182.84) | 2250.00 (821.30)

4. Secondary Outcome: Dose Normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast[dn])
Description: AUClast[dn] = Dose normalized area under the plasma concentration time-curve (AUC[dn]) from zero to the last measured concentration.
Time Frame: as for outcome 2
Population: PK parameter analysis population included all enrolled and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL/mg
Arm/Group | Crizotinib 50 mg IV | Crizotinib 250 mg Oral
Number analyzed (Participants) | 14 | 14
ng*hr/mL/mg | 20.14 (3.63) | 9.00 (3.28)
Statistical Analysis 1: Comparison: Crizotinib 50 mg IV vs Crizotinib 250 mg Oral; Natural log transformed AUClast(dn) of crizotinib was analyzed using mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences was exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 44.67, 90% CI 2-sided [40.90 to 48.78]

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Crizotinib 50 mg IV | Crizotinib 250 mg Oral
Number analyzed (Participants) | 14 | 14
ng/mL | 155.00 (29.57) | 99.60 (28.82)

6. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, and 144 hrs post oral crizotinib dose in Treatment B
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Crizotinib 250 mg Oral
Number analyzed (Participants) | 14
hr | 5.0 [4.0 to 6.0]

7. Secondary Outcome: Plasma Decay Half Life (t1/2)
Description: Plasma decay half life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Crizotinib 50 mg IV | Crizotinib 250 mg Oral
Number analyzed (Participants) | 14 | 14
hr | 38.86 (6.10) | 28.98 (2.96)

8. Secondary Outcome: Apparent Oral Clearance (CL/F)
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Time Frame: 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, and 144 hrs post oral crizotinib dose in Treatment B
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: L/hr
Arm/Group | Crizotinib 250 mg Oral
Number analyzed (Participants) | 14
L/hr | 107.7 (36.1)

9. Secondary Outcome: Systemic Clearance (CL)
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: 0 (pre-dose), 1, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 144 hrs post IV crizotinib dose in Treatment A
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: L/hr
Arm/Group | Crizotinib 50 mg IV
Number analyzed (Participants) | 14
L/hr | 46.83 (8.64)

10. Secondary Outcome: Apparent Volume of Distribution (Vz/F)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, and 144 hrs post oral crizotinib dose in Treatment B
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: L
Arm/Group | Crizotinib 250 mg Oral
Number analyzed (Participants) | 14
L | 4478.0 (1665.3)

11. Secondary Outcome: Volume of Distribution at Steady State (Vss)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.
Time Frame: 0 (pre-dose), 1, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 144 hrs post IV crizotinib dose in Treatment A
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: L
Arm/Group | Crizotinib 50 mg IV
Number analyzed (Participants) | 14
L | 1772.00 (328.75)

12. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for Crizotinib Metabolite (PF-06260182)
Description: Area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration (AUClast) of crizotinib metabolite (PF-06260182).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib 50 mg IV | Crizotinib 250 mg Oral
Number analyzed (Participants) | 14 | 14
ng*hr/mL | 35.61 (17.64) | 342.70 (116.22)

13. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC [0 - ∞]) for Crizotinib Metabolite (PF-06260182)
Description: AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞) of crizotinib metabolite (PF-06260182).
Time Frame: 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, and 144 hrs post oral crizotinib dose in Treatment B
Population: PK parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period. Here, the 'N = 13' is signifying those participants who were evaluable for this measure at the specified time point for this arm group.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib 250 mg Oral
Number analyzed (Participants) | 13
ng*hr/mL | 360.4 (117.2)

14. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Crizotinib Metabolite (PF-06260182)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Crizotinib 50 mg IV | Crizotinib 250 mg Oral
Number analyzed (Participants) | 14 | 14
ng/mL | 3.01 (1.46) | 26.46 (6.41)

15. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for Crizotinib Metabolite (PF-06260182)
Time Frame: 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, and 144 hrs post oral crizotinib dose in Treatment B
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Crizotinib 250 mg Oral
Number analyzed (Participants) | 14
hr | 5.00 [5.00 to 6.07]

16. Secondary Outcome: Metabolite to Parent Ratio of Area Under the Curve From Time Zero to Last Quantifiable Concentration for Crizotinib Metabolite Ratio (MRAUClast)
Description: Molar ratio of metabolite to parent area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration (MRAUClast).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Crizotinib 50 mg IV | Crizotinib 250 mg Oral
Number analyzed (Participants) | 14 | 14
Ratio | 0.034 (0.011) | 0.148 (0.021)

17. Secondary Outcome: Metabolite to Parent Ratio Area Under the Curve From Time Zero to Extrapolated Infinite Time (MRAUC [0-∞])
Description: Molar ratio of metabolite to parent area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-∞) (MRAUC [0-∞]).
Time Frame: 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, and 144 hrs post oral crizotinib dose in Treatment B
Population: as for outcome 13
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Crizotinib 250 mg Oral
Number analyzed (Participants) | 13
Ratio | 0.144 (0.019)

18. Secondary Outcome: Metabolite to Parent Ratio Maximum Observed Plasma Concentration (MRCmax)
Description: Metabolite to parent molar ratio of maximum observed plasma concentration (MRCmax).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Crizotinib 50 mg IV | Crizotinib 250 mg Oral
Number analyzed (Participants) | 14 | 14
Ratio | 0.019 (0.007) | 0.258 (0.043)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Crizotinib 50 mg IV | Crizotinib 250 mg Oral
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 8/14 | 5/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crizotinib 50 mg IV (N=14) | Crizotinib 250 mg Oral (N=14)
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Flatulence (Gastrointestinal disorders) | 1 | 1
Catheter site pain (General disorders) | 2 | 0
Catheter site phlebitis (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes